CLINICAL TRIAL: NCT06274294
Title: The "PASSPORT Trial": Pharmacokinetics, Efficacy and Safety of CT-P13 Subcutaneous as Induction Therapy in Patients With Active Crohn's Disease or Ulcerative Colitis.
Brief Title: Pharmacokinetics, Efficacy and Safety of CT-P13 Subcutaneous as Induction Therapy in Patients With Active CD or UC
Acronym: PASSPORT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CMC Ambroise Paré (Other)
Collaborators: Paris IBD Center (Other); Celltrion HealthCare France (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/12
Record Dates: First submitted 2024-02-07; First posted 2024-02-23 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-02

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Inflammatory Bowel Diseases; Crohn's disease; Ulcerative colitis; Infliximab / CT-P13; Intravenous; Subcutaneous; Pharmacokinetics; Efficacy; Safety; AUC; Ctrough; Fecal calprotectin; Antibodies to infliximab; C-reactive protein; TSQM; IBD disability index
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — CT-P13

STUDY DESIGN:
Intervention Model Description: The full sample size comprises 130 patients, with 65 patients allocated to each arm. The arms are defined as follows:
  * Experimental Arm: Patients receive CT-P13 SC at weeks 0, 1, 2, 3, 4, and 6, followed by subcutaneous administration every two weeks until week 24.
  * Control Arm: Patients receive CT-P13 IV at weeks 0 and 2, followed by subcutaneous administration every two weeks until week 24.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SC CT-P13 induction (Experimental): Experimental arm: SC induction of 240 mg of CT-P13 at week 1, then 120 mg at weeks 2, 3, 4 then every 2 weeks until week 24.
  Interventions: Drug: CT-P13
- IV CT-P13 induction (Other): Control arm: IV induction of 5 mg/kg of CT-P13 at weeks 1 and 2 then SC (120 mg) every 2 weeks until week 24.
  Interventions: Drug: CT-P13

INTERVENTIONS:
Drug: CT-P13 — Induction treatment.

SUMMARY:
The goal of this clinical trial is to compare induction treatment with CT-P13 SC to induction treatment with CT-P13 IV in terms of pharmacokinetics in adult patients with inflammatory bowel disease (IBD) who have been diagnosed for at least 3 months and for whom the physician has decided to initiate treatment with infliximab CT-P13 as part of the standard of care.

The main aim of this study is to demonstrate that induction treatment with CT-P13 SC is non-inferior to CT-P13 IV in terms of pharmacokinetics at Week 6.

DETAILED DESCRIPTION:
The subcutaneaous formulation of infliximab CT-P13 represents a promising approach in the treatment of inflammatory bowel disease (IBD), with an efficacy/safety/immunogenicity profile similar or even improved compared to the intravenous formulation of CT-P13. For patients, SC administration can offer benefits over their daily activities by reducing the frequency of days spent in the hospital to receive infusions. The SC administration may offer convenience for the healthcare system, optimizing the organizational impact due to the preparation and administration of the IV infusion, allowing resources to be used more efficiently, and reducing direct costs associated with the infusion. There are no clinical trials with Remsima® 120 mg given subcutaneously without IV loading doses of CT-P13 in patients with IBD. However, population pharmacokinetic and pharmacokinetic/pharmacodynamic modelling and simulation predicted comparable CT-P13 exposure (AUC over 8 weeks) and efficacy from Week 6 onward in rheumatoid arthritis patients treated with Remsima® 120 mg given without IV loading doses of CT-P13 when compared with Remsima® 3 mg/kg given intravenously at weeks 0, 2 and 6, and then every 8 weeks. For the dosing regimen with subcutaneous loading in patients with rheumatoid arthritis, the predicted median AUC value was 17,400 μg·h/mL from Week 0 to 6 which was approximately 1.8 fold lower than the predicted median AUC value for the dosing regimen with CT-P13 IV loading doses (32,100 μg·h/mL). Whereas the predicted median AUC values from Week 6 to 14 were comparable between the two dosing regimens with SC loading and IV loading (19,600 and 18,100 μg·h/mL, respectively).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged at least 18 years old.
2. Diagnosis of inflammatory bowel disease according to the ECCO criteria for at least 3 months:

   * moderately to severely active CD (Crohn's disease)
   * moderately to severely active UC (Ulcerative colitis)
3. Patients had received conventional therapy for active UC (corticosteroids alone or in combination with thiopurines and 5-aminosalicylates) or CD (corticosteroids and/or immunomodulators) but had not responded despite an adequate course of therapy.
4. Patient has active CD or UC with at least one objective sign of disease activity on biology, endoscopy or imaging.
5. Initiation of infliximab CT-P13 as part of standard of care.
6. Patient suffering from anal suppuration related to CD can be included.
7. Person who has received full information about the organization of the research, who has not objected to his or her participation and to the use of his or her data.
8. Person affiliated to or beneficiary of a social security plan.
9. ► Inclusion criteria for Women of Childbearing Age:

Women of childbearing age should consider the use of appropriate contraception to prevent pregnancy and continue its use for at least 6 months after the last infliximab treatment. Women should choose one of the following methods of contraception:

* Combined hormonal contraception containing estrogen and progesterone (oral, IUD, transdermal, injectable) combined with ovulation inhibition.
* Initiated at least 30 days before Baseline Day 1.
* Progestin-only hormonal contraception (oral, injectable, implantable) associated with ovulation inhibition initiated at least 30 days before the first injection.
* Bilateral tubal occlusion (can be performed by hysteroscopy, provided that hysterosalpingography confirms the success of the procedure).
* Intrauterine device (IUD).
* Practicing true abstinence, defined as: abstaining from heterosexual intercourse when this corresponds to the subject's preferred and usual lifestyle (periodic abstinence [e.g. calendar method, ovulation method, symptothermal method, post-ovulation methods] and withdrawal are not acceptable)

  * Inclusion Criteria for Women Not of Childbearing Age:

Women do not need to use contraception during or after treatment with study drug if they are considered not of childbearing age due to one of the following situations:

* Premenopausal women with permanent infertility following hysterectomy, bilateral salpingectomy or bilateral oophorectomy.
* Postmenopausal women
* Age > 55 years without menstruation for 12 months or more without alternative medical cause.
* Age ≤ 55 years without menstruation for 12 months or more without alternative medical cause AND a folliculostimulin (FSH) level > 30 IU/L.

Exclusion Criteria:

1. Combination therapy with an immunomodulator except for patients suffering from anal suppuration related to CD.
2. Patient who has allergies to any of the excipients of infliximab CT-P13 or any other murine and/or human proteins or patient with a hypersensitivity to immunoglobulin product.
3. Patient who had current or past history of chronic infection with hepatitis C or human immunodeficiency virus (HIV)-1 or -2 or current infection with hepatitis B.
4. Patient who had acute infection requiring oral antibiotics within 2 weeks or parenteral injection of antibiotics within 4 weeks prior to the first administration of the study drug, other serious infection within 6 months prior to the first administration of study drug or recurrent herpes zoster or other chronic or recurrent infection within 6 weeks prior to the first administration of the study drug.
5. Patients with a positive interferon-γ release assay (IGRA) or latent tuberculosis (TB) prior to initiation of biologic therapy.
6. Patients with moderate or severe heart failure (NYHA class III/IV).
7. Person referred in articles L.1121-5, L. 1121-7 and L.1121-8 of the Public Health Code: pregnant woman, parturient, or breastfeeding woman, minor person (non-emancipated), adult person under legal protection (any form of public guardianship), adult person incapable of giving consent.
8. Person deprived of liberty for judicial or administrative decision, person under psychiatric care as referred in articles L. 3212-1 and L. 3213-1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Ratio SC/IV | Week 6
  The ratio (SC/IV) of log-normal means of Ctrough at W6 and its 95% CI. Non inferiority will be considered as demonstrated if the lower limit of the 95%CI is higher than 80%.

SECONDARY OUTCOMES:
Ctrough at week 24 (non-inferiority) | Week 24
AUC at week 24 | Week 24
Clinical response at week 6 and week 24 | Weeks 6 and 24
  * Defined for UC as a decrease of at least 50% in PRO2.
  * Defined for CD as a decrease from baseline in CDAI score of at least 100 points or a total CDAI score < 150 and defined as achieving a total HBI < 4
IBD disability index at week 6 | Week 6
Fecal calprotectin at week 24 | Week 24
Clinical remission at week 6 and week 24 | Weeks 6 and 24
  * Defined for UC as a symptomatic remission score with a stool frequency subscore of 0 or a subscore of 1 with a decrease of ≥1 point from baseline, and a rectal-bleeding subscore of 0.
  * Defined for CD as a CDAI score < 150 evaluated in semi-blind (assessment will be done by another investigator without information on the treatment) and defined as achieving a total HBI < 4.
Presence of antibodies to infliximab at Week 6 and Week 24 | Weeks 6 and 24
Concentration of C-reactive protein up to week 6 (the samples are collected at weeks 0, 6 and 24) | Up to Week 6
Adverse events, including injection site reactions and hypersensitivity reactions | From Baseline up to 6 weeks and 24 weeks
  Number of participants, number of AEs per patient, number of injection site reactions and hypersensitivity reactions per patient.
TSQM collected at Week 6 and Week 24 | 24 months
  The Treatment Satisfaction Questionnaire for Medication consists of 14 items that results in four specific domains: Effectiveness, Side Effects, Convenience, and one global scale item, Global Satisfaction. Scores for each domain are computed by adding the TSQM items in each domain and then transforming the composite score into a value ranging from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Bouhnik, PhD.Med., Principal Investigator — Paris IBD Center
Locations (1):
- Institut des MICI, Neuilly-sur-Seine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schreiber S, Ben-Horin S, Leszczyszyn J, Dudkowiak R, Lahat A, Gawdis-Wojnarska B, Pukitis A, Horynski M, Farkas K, Kierkus J, Kowalski M, Lee SJ, Kim SH, Suh JH, Kim MR, Lee SG, Ye BD, Reinisch W. Randomized Controlled Trial: Subcutaneous vs Intravenous Infliximab CT-P13 Maintenance in Inflammatory Bowel Disease. Gastroenterology. 2021 Jun;160(7):2340-2353. doi: 10.1053/j.gastro.2021.02.068. Epub 2021 Mar 5. PMID 33676969
- [Result] Iannone F, Conti F, Cauli A, Farina A, Caporali R. Subcutaneously-Administered Infliximab in the Management of Rheumatoid Arthritis: A Short Narrative Review of Current Clinical Evidence. J Inflamm Res. 2022 Jun 1;15:3259-3267. doi: 10.2147/JIR.S240593. eCollection 2022. PMID 35673354